CLINICAL TRIAL: NCT03667703
Title: Stress Ulcer Prophylaxis Versus Placebo - a Blinded Randomized Control Trial to Evaluate the Safety of Two Strategies in Critically Ill Infants With Congenital Heart Disease
Brief Title: Stress Ulcer Prophylaxis Versus Placebo in Critically Ill Infants With Congenital Heart Disease
Acronym: SUPPRESS-CHD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Collaborators: The Gerber Foundation (Other)
Responsible Party: Principal Investigator, Kimberly I. Mills, MD, Assistant in Cardiology, Instructor in Pediatrics, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: IRB-P00028715
Record Dates: First submitted 2018-07-13; First posted 2018-09-12 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Congenital Heart Disease; Upper Gastrointestinal Bleeding; Stress Ulcer; Infection
MeSH Terms: conditions — Heart Defects, Congenital; Gastrointestinal Hemorrhage; Duodenal Ulcer; Infections | interventions — Famotidine; Saline Solution

STUDY DESIGN:
Intervention Model Description: Prospective, double-blinded randomized placebo-controlled pilot feasibility trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): Subjects randomized to placebo will receive an equivalent volume (mL) of normal saline intravenously or Ora-plus orally based on weight and age.
  Interventions: Drug: Placebo
- Study Drug (Active Comparator): Subjects randomized to study drug will receive famotidine, a histamine-2 receptor antagonist. Dosing will be weight based and age-dependent. Infants < 90 days old will receive either 0.5mg/kg intravenously daily or 0.5mg/kg orally twice a day of famotidine. Infants ≥ 90 days or older will receive 0.25mg/kg intravenously every 12 hours or 0.5mg/kg orally twice a day.
  Interventions: Drug: Famotidine

INTERVENTIONS:
Drug: Famotidine — Patients will be randomized to either receive a placebo or famotidine (study drug).
  Other Names: Pepcid
  Arms: Study Drug
Drug: Placebo — Patients will be randomized to either receive a placebo or famotidine (study drug).
  Other Names: Normal saline or stevoside-free syrup
  Arms: Placebo

SUMMARY:
Infants with congenital heart disease often require an intervention during their first year of life. Infants are generally admitted to a cardiac intensive care unit and are routinely prescribed stress ulcer prophylaxis to decrease acid release from the stomach to prevent stress ulcer formation. However, these medicines may not be safe and could put infants at increased risk for hospital-acquired infections, necrotizing enterocolitis and alteration to the infant's microbiome. The investigators plan to assess the feasibility of conducting a prospective, blinded randomized control trial to determine the safety of withholding stress ulcer prophylaxis in critically ill infants with congenital heart disease. In addition, the investigators plan to examine the changes to the infant's microbiome through oral, gastric and stool samples and compare hospital-acquired infections.

DETAILED DESCRIPTION:
Background & Significance. Approximately 36,000 infants are born with congenital heart disease (CHD) in the United States each year, often requiring surgical intervention in the first year of life. They are vulnerable to postoperative morbidities including infection, growth failure and neurodevelopmental delay. Upon admission to the cardiac intensive care unit (CICU), infants are routinely prescribed stress ulcer prophylaxis (SUP) to decrease acid release from the stomach thus preventing ulcer-induced upper gastrointestinal (UGI) bleeding. Although adopted from the adult literature, this practice is expensive and has not been shown to be effective in infants. More importantly, recent literature suggests that this may not be safe. Studies show an increased risk of hospital-acquired infections, necrotizing enterocolitis and alterations in the evolving healthy gut flora in infants. The study investigators have recently demonstrated an increased risk of infection in children receiving SUP and also reported differences in microbial diversity among children in the CICU. It is necessary to proceed with a prospective trial to determine the safety of withholding SUP in critically ill children with CHD.

Specific Aims & Hypothesis. The overarching hypothesis of the proposal is withholding SUP from critically ill infants with CHD is safe and results in favorable microbial diversity, thus decreasing hospital-acquired infections. Primary Aim 1 of the study is to assess the feasibility of this pilot randomized, controlled clinical trial of SUP versus placebo in infants admitted to the CICU. The study investigators hypothesize that a priori feasibility measures will be achieved during the study period. Primary Aim 2 of the study is to examine the differences of UGI bleeding in critically ill infants with CHD receiving SUP versus those receiving placebo. The study investigators hypothesize that the rate of UGI bleeding will be no different between infants exposed to SUP and to placebo. Secondary Aim 1 of the study is to compare the differences in the abundance of microbial taxa and functional profiles of the aerodigestive tract microbiome between infants receiving SUP and those receiving placebo and before/after the start of SUP. The study investigators hypothesize that there will be significant differences in the abundance of microbial taxa and the functional profiles between the 2 groups - with a more favorable microbial profile present in infants in the placebo group. Secondary Aim 2 is to examine the difference in the incidence of hospital-acquired infections in critically ill infants with CHD receiving SUP versus placebo. The study investigators hypothesize the rate of hospital-acquired infections will be higher in patients exposed to SUP when compared to placebo.

Study Design & Methods. A single-center, prospective, double-blinded, randomized, controlled trial will be conducted as a feasibility study for a larger multicenter trial. Consecutive infants < 12 months of age with CHD admitted to the CICU and anticipated to require respiratory support for > 24 hours will be enrolled and randomized to receive a histamine-2 receptor antagonist (H2RA) medication or study placebo. Patients will remain in the study until discontinuation of respiratory support, discharge from the CICU or study day 14. Oral, gastric and stool samples will be obtained prior to receiving the first dose of study drug and subsequently at the end of the study. The samples will be analyzed for 16S RNA and metagenomic shotgun sequencing for microbiome composition. Gastric pH will be recorded on all gastric samples. Demographics, nutrition variables, medications, and respiratory data will be collected for all patients while enrolled in the study. An independent Drug Safety and Monitoring Board (DSMB) will monitor patient safety every 6 months and after any significant adverse event.

Outcomes. The primary outcomes will be study feasibility and incidence of clinically significant UGI bleeding. Feasibility will be defined as: 1) > 80% screening of eligible patients, 2) > 20% consent rate, 3) > 80% receive timely first dose of study drug, and 4) > 80% protocol adherence. Clinically significant UGI bleeding will be defined as new-onset bleeding with subsequent pre-defined physiologic or hemodynamic changes. The secondary outcomes of the study will be observed differences in the aerodigestive microbial diversity between study groups, mortality, length of stay, duration of respiratory support, bleeding events, incidence of necrotizing enterocolitis and incidence of hospital-acquired infections (ventilator-associated pneumonia, central line-associated bloodstream infections, catheter-associated urinary tract infections, superficial sternal infection or mediastinitis).

ELIGIBILITY:
Inclusion Criteria:

1. < 12 months of age (including premature newborns),
2. diagnosed with congenital heart disease (including anatomic, myopathic and arrhythmic conditions),
3. received ≤ 1 dose of SUP (including histamine-2 receptor antagonists, proton pump inhibitors, and sucralfate) during current admission, AND
4. anticipated to require respiratory support for > 24 hours during their CICU stay. Respiratory support includes mechanical ventilation, non-invasive positive-pressure ventilation and high-flow oxygen therapy.

Exclusion Criteria:

1. prior use of antacids (including histamine-2 receptor antagonists, proton pump inhibitors, or sucralfate) in the past month for > 7 days,
2. active gastrointestinal bleeding,
3. active Helicobacter pylori infection,
4. administration of high-dose steroids (equivalent dosing to 15 mg/kg/day of methylprednisolone),
5. will receive ketorolac (intravenous nonsteroidal anti-inflammatory drug) during admission,
6. exposed to specific anticoagulants (high-dose aspirin, direct thrombin inhibitors and GPIIbIIIa inhibitors),
7. planned to undergo or recently has undergone gastrointestinal surgery (i.e. repair of duodenal atresia)
8. supported by extracorporeal membrane oxygenator (ECMO) or ventricular assist device (VAD),
9. currently enrolled in another intervention trial,
10. known to be allergic to H2RAs,
11. admitted for palliative care,
12. prior enrollment in the study, OR
13. primary provider declines enrollment.

Ages: 1 Minute to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 70 (Actual)
Dates: Start 2019-03-10 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Predefined Feasibility Outcomes to Assess Trial Success | Through study completion, anticipated 2 years.
  Feasibility will be defined by the following metrics: (1) if >80% of eligible patients are approached for consent (screening), (2) >20% of eligible patients are randomized (consent and enrollment), (3) >80% of enrolled patients received first dose of study drug within 48 hours (allocation), and (4) >80% compliance to protocol and treatment group (protocol adherence).
Rate of upper gastrointestinal bleeds | Through study completion, anticipated 2 years.
  To examine the difference in the incidence of clinically significant upper gastrointestinal (UGI) bleeding in critically ill infants with CHD receiving SUP versus placebo to demonstrate safety.

SECONDARY OUTCOMES:
Microbiome alterations | Through study completion, anticipated 2 years.
  To compare the absolute and serial differences in the abundance of bacteria and functional microbial profiles in the aerodigestive tract between critically ill infants with CHD receiving SUP compared to placebo.
Rate of hospital-acquired infections | Through study completion, anticipated 2 years.
  To examine the difference in the incidence of hospital-acquired infections in critically ill infants with CHD receiving SUP versus placebo. Hospital-acquired infections include ventilator-associated pneumonia, central line-associated bloodstream infections, catheter-associated urinary tract infections, superficial sternal infection, or mediastinitis.

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly I Mills, MD, Principal Investigator — Boston Children's Hospital; Ben D Albert, MD, Principal Investigator — Boston Children's Hospital; Nilesh M Mehta, MD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mills KI, Albert BD, Bechard LJ, Chu S, Duggan CP, Kaza A, Rakoff-Nahoum S, Sleeper LA, Newburger JW, Priebe GP, Mehta NM. Stress Ulcer Prophylaxis Versus Placebo-A Blinded Pilot Randomized Controlled Trial to Evaluate the Safety of Two Strategies in Critically Ill Infants With Congenital Heart Disease. Pediatr Crit Care Med. 2024 Feb 1;25(2):118-127. doi: 10.1097/PCC.0000000000003384. Epub 2024 Jan 19. PMID 38240536
- [Derived] Mills KI, Albert BD, Bechard LJ, Duggan CP, Kaza A, Rakoff-Nahoum S, Vlamakis H, Sleeper LA, Newburger JW, Priebe GP, Mehta NM. Stress ulcer prophylaxis versus placebo-a blinded randomized control trial to evaluate the safety of two strategies in critically ill infants with congenital heart disease (SUPPRESS-CHD). Trials. 2020 Jun 29;21(1):590. doi: 10.1186/s13063-020-04513-w. PMID 32600393